CLINICAL TRIAL: NCT00138684
Title: Cytochrome P450 2E1 and Iron Overload
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DGS 2003/0052; PHRC/02-09 (Other: Rennes University Hospital); CIC0203/015
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Insulin Resistance; Iron Overload
Keywords: insulin resistance; iron overload; phlebotomy; hepatic iron overload
MeSH Terms: conditions — Insulin Resistance; Iron Overload | interventions — Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Venesection therapy (Experimental)
  Interventions: Procedure: venesection
- no venesection therapy (No Intervention)

INTERVENTIONS:
Procedure: venesection — Venesection therapy is realised every 7 - 14 days until iron desaturation completion.
  Arms: Venesection therapy

SUMMARY:
The aim of the study is to determine, in patients presenting hepatic iron overload (genetic haemochtomatisis or dysmetabolic iron overload syndrome), the effects of venesection therapy on cytochrome P450 2E1 activity by comparing the rates of metabolization of chlorzoxazone before and after venesection.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged from 18 to 70 years
* Hepatic iron overload measured by magnetic resonance imaging [MRI] (> 36 µmol/g and < 200 µmol/L)
* Homozygosity for the C282Y mutation of the HFE or dysmetabolic iron overload syndrome (DIOS) based on the presence of at least one of these following metabolic abnormalities:
* Overweight: BMI > 25 kg/m2
* Waist/hip circumference (cm) > 0.90
* Diabetes mellitus (fasting blood glucose level >1.25g/L or blood glucose level after 2 hours > 2g/L) or glucose intolerance (fasting blood glucose level between 1.10 and 1.25g/L)
* Total cholesterolemia > 6.2 mmol/L or HDL-Cholesterol < 0.9 mmol/L
* TG>= 1.7 mmol
* Written informed consent

Non-Inclusion Criteria:

* Consumption of alcohol > 50 g/day and of any CYP2E1 inhibitor substances
* Smoker > 5 cigarets/day
* History of blood donation or venesection
* Other causes of iron overload: aceruloplasminaemia, haematological disorder (abnormal blood counting), late cutaneous porphyria (cutaneous bullous disorders and photosensibilisation) , martial treatment, repeated transfusions.
* Inflammatory syndrome (CRP > 3ng/ml)

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-09; Primary Completion 2005-12 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
variation of chlorzoxazone metabolization rate measured before and after venesection | Baseline and after iron desaturation completion

SECONDARY OUTCOMES:
variation of blood Malonedialdehyde rate | Baseline and after iron desaturation completion
variation of blood 4-hydroxynonenal rate | Baseline and after iron desaturation completion
variation of blood Glutathion rate | Baseline and after iron desaturation completion
variation of serum Vitamin E rate | Baseline and after iron desaturation completion
Variation of serum Vitamin C rate | Baseline and after iron desaturation completion

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Reymann, PhD, Study Chair — CHU Rennes; Fabrice Lainé, MD, Principal Investigator — CHU Rennes
Locations (2):
- France (2):
  - CHU Nantes, Nantes
  - Unité d'Investigation Clinique - Hôpital Pontchaillou, Rennes